CLINICAL TRIAL: NCT06500468
Title: Usage of Novel Blood Sensing Capsule in Emergency Department to Triage Patients With Suspected Upper Gastrointestinal Bleeding
Brief Title: PillSense for Suspected Upper Gastrointestinal Bleeding
Acronym: BLEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: EnteraSense Limited (Industry)
Responsible Party: Principal Investigator, Wee Khoon Ng, Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/00060
Record Dates: First submitted 2024-07-06; First posted 2024-07-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Bleeding Ugi
Keywords: capsule endoscopy; upper gastrointestinal bleeding; melena; coffee ground vomitting; emergency department; triage
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Melena; Emergencies

STUDY DESIGN:
Intervention Model Description: Partipants will be randomised into either of the 2 arms: PillSense Group (Treatment arm) or Standard group (where they will receive standard of care) for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PillSense group (Experimental): Participants in the PillSense arm will swallow one PillSense capsule. Participants who have blood detected will be admitted with a scheduled oesophagogastroduodenoscopy within 72 hours. Participants with no blood detected will be discharged with medications and a scheduled OGD within 96 hours.
  Interventions: Device: PillSense System
- Standard group (No Intervention): Participants randomized to the standard arm will follow standard of care and will either be admitted or discharged with medications and to undergo an oesophagogastroduodenoscopy (OGD) within 72 hours if admitted or 96 hours if discharged.

INTERVENTIONS:
Device: PillSense System — The PillSense System consists of the PillSense Capsule, a small single use capsule that is safe for human consumption and PillSense Receiver, an external real-time monitor for data display. The PillSense Capsule is a minimally invasive, single use medical device designed to detect the presence of bleeding in the upper digestive tract, to aid with patient care. The PillSense Receiver collects and displays real-time information gathered by the PillSense Capsule within 10 minutes. The PillSense Receiver interprets the data and displays a result message "Blood detected" or "No blood detected".
  Arms: PillSense group

SUMMARY:
This study aims to evaluate the efficacy and safety of a novel blood sensing capsule (PillSense), to help emergency doctors better evaluate if patients have active upper digestive tract bleeding, to determine if they can be discharged safely. The PillSense System consists of the PillSense Capsule, a small single use capsule that is safe for human consumption and PillSense Receiver, an external real-time monitor for data display to detect the presence of bleeding in the upper digestive tract within 10 minutes.

DETAILED DESCRIPTION:
The use of the PillSense System enables the clinician to make a more informed choice on the treatment plan for the patient. If the system revealed "No Blood Detected", this is suggestive there is absence of blood in the stomach. Together with the presenting symptoms, physical examination and laboratory tests, it gives the emergency physician a more accurate method to detect if patient is actively bleeding. If patient remained stable during the monitoring, the patient can be discharged home for early outpatient review, instead of waiting in Emergency Department (ED) for prolonged duration to be admitted and wait in the ward for investigations like gastroscopy to be performed. This reduces unnecessary strain on the hospital's limited resources and may improve overall patient's experience. Patients with 'Blood Detected' result will be admitted with early gastroscopy planned within 72 hours. Patients with 'No Blood Detected' result, will be monitored closely in ED and, if deemed to be stable, to be discharged with an outpatient gastroscopy within 96 hours. A product such as the PillSense System which employs a minimally invasive method to help clinicians detect whether or not a patient has blood in upper gastrointestinal tract within 10 minutes. This will be a quick and objective tool to determine if the patient is having active upper gastrointestinal bleeding (UGIB), to assist in triaging patients for more emergent definitive care. This system can also be easily administered by non-clinician and do not require special training to read the results, minimising the need for highly specialised staff to provide this service. The information provided by the PillSense System which taken together with other clinical parameters may lead to more efficient, safer and higher quality patient care.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 21 years and above and are able to give consent.
* Patients who are willing and able to comply with the study protocol (including undergoing endoscopy)
* Presented to Emergency Department with symptoms of acute overt upper gastrointestinal bleeding such as coffee ground vomiting and melena (but without melaena on physical examination)

Exclusion Criteria:

* Patients who had hemodynamic shock (systolic blood pressure below 90 mm Hg and pulse rate over 120/min)
* Patients who presented with fresh hematemesis, hematochezia and/or melaena
* Patients requiring urgent endoscopy / surgery at time of review or already planned for admission by ED physician for non UGIB related indications
* Patients who had conditions that might contraindicate the use of an ingestible capsule, such as capsule endoscopy (eg. Dysphagia, odynophagia, swallowing disorder, and/or Zenker's diverticulum, issues with the motility of the gastrointestinal tract, Crohn's disease, previous GI surgery, suspected ileus, bowel obstruction and/or perforation)
* Patients with a known history of oesophageal or gastric varices
* Patients with known UGI pathology (such as oesophageal/gastric cancer), or recent (within 3 months) upper GI ulcer bleeding, upper GI surgeries or procedures
* Patients who are on anticoagulation
* Patients with cardiac implantable electrical device (CIED)
* Patients who had altered mental status
* Pregnant and/or lactating women (Female patients below age 60, without history of hysterectomy or are not documented to be post-menopausal, will be given a urine pregnancy test to confirm they are not pregnant)
* Patients who have an MRI investigation planned within 2 weeks

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Discharge rate of patients with stable UGIB who can be triaged home safely after ED visit | 1.5 years
  To compare the percentage of patients who are safely discharged from ED visit with the usage of PillSense, compared to standard treatment.

SECONDARY OUTCOMES:
Risk of clinical rebleeding after a negative PillSense reading | 1.5 years
  To measure the number of patients who have clinical re-bleeding in both arms.
Discharge rate of patients who can be triaged home using PillSense , compared to conventional clinical scoring system like Glasgow Blatchford Score (GBS). | 1.5 years
  To compare what is the percentage of patients who can be discharged safely using PillSense vs Glasgow Blatchford Score alone. The Glasgow Blatchford Score (GBS) is a risk assessment tool to help triage patients presenting with upper gastrointestinal bleeding, if they can be discharged safely from emergency department for outpatient care. The score may range from 0 to 23 and higher scores are associated with higher risks of complications related to gastrointestinal bleeding. Conventional studies recommend that such patients can be safely discharged if the score is 0.
Number of inpatient beds saved from this arrangement | 1.5 years
  To review the beds and potential cost savings from the hospital from the reduction of admissions
Risk of patient morbidity after a negative PillSense reading | 1.5 years
  To quantify and specify any patient morbidity after a negative PillSense reading.
Risk of patient mortality after a negative PillSense reading | 1.5 years
  To quantify and specify any mortality after a negative PillSense reading.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ng Wee Khoon, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gleeson F, Clarke E, Lennon J, MacMathuna R, Crowe J. Outcome of accident and emergency room triaged patients with low risk non-variceal upper gastrointestinal haemorrhage. Ir Med J. 2006 Apr;99(4):114-7. PMID 16972584
- [Background] Owensby S, Taylor K, Wilkins T. Diagnosis and management of upper gastrointestinal bleeding in children. J Am Board Fam Med. 2015 Jan-Feb;28(1):134-45. doi: 10.3122/jabfm.2015.01.140153. PMID 25567834
- [Background] Biecker E, Heller J, Schmitz V, Lammert F, Sauerbruch T. Diagnosis and management of upper gastrointestinal bleeding. Dtsch Arztebl Int. 2008 Feb;105(5):85-94. doi: 10.3238/arztebl.2008.0085. Epub 2008 Feb 1. PMID 19633792
- [Background] Ferguson CB, Mitchell RM. Non-variceal upper gastrointestinal bleeding. Ulster Med J. 2006 Jan;75(1):32-9. No abstract available. PMID 16457402
- [Background] Rockall TA, Logan RF, Devlin HB, Northfield TC. Incidence of and mortality from acute upper gastrointestinal haemorrhage in the United Kingdom. Steering Committee and members of the National Audit of Acute Upper Gastrointestinal Haemorrhage. BMJ. 1995 Jul 22;311(6999):222-6. doi: 10.1136/bmj.311.6999.222. PMID 7627034
- [Background] Rockall TA, Logan RF, Devlin HB, Northfield TC. Risk assessment after acute upper gastrointestinal haemorrhage. Gut. 1996 Mar;38(3):316-21. doi: 10.1136/gut.38.3.316. PMID 8675081
- [Background] Zimmerman J, Meroz Y, Arnon R, Tsvang E, Siguencia J. Predictors of mortality in hospitalized patients with secondary upper gastrointestinal haemorrhage. J Intern Med. 1995 Mar;237(3):331-7. doi: 10.1111/j.1365-2796.1995.tb01183.x. PMID 7891055
- [Background] Schembre DB, Ely RE, Connolly JM, Padhya KT, Sharda R, Brandabur JJ. Semiautomated Glasgow-Blatchford Bleeding Score helps direct bed placement for patients with upper gastrointestinal bleeding. BMJ Open Gastroenterol. 2020 Nov;7(1):e000479. doi: 10.1136/bmjgast-2020-000479. PMID 33214231
- [Background] Fisher L, Fisher A, Pavli P, Davis M. Perioperative acute upper gastrointestinal haemorrhage in older patients with hip fracture: incidence, risk factors and prevention. Aliment Pharmacol Ther. 2007 Feb 1;25(3):297-308. doi: 10.1111/j.1365-2036.2006.03187.x. Epub 2007 Jan 8. PMID 17217452
- [Background] Sengupta N. Integrating Gastrointestinal Bleeding Risk Scores into Clinical Practice. Am J Gastroenterol. 2019 Nov;114(11):1699-1703. doi: 10.14309/ajg.0000000000000417. No abstract available. PMID 31592783
- [Background] Sachdev MS, Leighton JA, Fleischer DE, Heigh RI, Hara AK, Post JA, Erickson PJ, Sharma VK. A prospective study of the utility of abdominal radiographs after capsule endoscopy for the diagnosis of capsule retention. Gastrointest Endosc. 2007 Nov;66(5):894-900. doi: 10.1016/j.gie.2007.06.066. PMID 17963875
- [Background] Rezapour M, Amadi C, Gerson LB. Retention associated with video capsule endoscopy: systematic review and meta-analysis. Gastrointest Endosc. 2017 Jun;85(6):1157-1168.e2. doi: 10.1016/j.gie.2016.12.024. Epub 2017 Jan 6. PMID 28069475
- [Background] Fernandez-Urien I, Carretero C, Gonzalez B, Pons V, Caunedo A, Valle J, Redondo-Cerezo E, Lopez-Higueras A, Valdes M, Menchen P, Fernandez P, Munoz-Navas M, Jimenez J, Herrerias JM. Incidence, clinical outcomes, and therapeutic approaches of capsule endoscopy-related adverse events in a large study population. Rev Esp Enferm Dig. 2015 Dec;107(12):745-52. doi: 10.17235/reed.2015.3820/2015. PMID 26671587
- [Background] Liao Z, Gao R, Xu C, Li ZS. Indications and detection, completion, and retention rates of small-bowel capsule endoscopy: a systematic review. Gastrointest Endosc. 2010 Feb;71(2):280-6. doi: 10.1016/j.gie.2009.09.031. PMID 20152309
- [Background] Lim YJ, Lee OY, Jeen YT, Lim CY, Cheung DY, Cheon JH, Ye BD, Song HJ, Kim JS, Do JH, Lee KJ, Shim KN, Chang DK, Park CH, Jang BI, Moon JS, Chun HJ, Choi MG, Kim JO; Korean Gut Image Study Group. Indications for Detection, Completion, and Retention Rates of Small Bowel Capsule Endoscopy Based on the 10-Year Data from the Korean Capsule Endoscopy Registry. Clin Endosc. 2015 Sep;48(5):399-404. doi: 10.5946/ce.2015.48.5.399. Epub 2015 Sep 30. PMID 26473123
- [Background] Rondonotti E, Soncini M, Girelli C, Ballardini G, Bianchi G, Brunati S, Centenara L, Cesari P, Cortelezzi C, Curioni S, Gozzini C, Gullotta R, Lazzaroni M, Maino M, Mandelli G, Mantovani N, Morandi E, Pansoni C, Piubello W, Putignano R, Schalling R, Tatarella M, Villa F, Vitagliano P, Russo A, Conte D, Masci E, de Franchis R; AIGO, SIED and SIGE Lombardia. Small bowel capsule endoscopy in clinical practice: a multicenter 7-year survey. Eur J Gastroenterol Hepatol. 2010 Nov;22(11):1380-6. doi: 10.1097/MEG.0b013e3283352ced. PMID 20173646
- [Background] Nemeth A, Wurm Johansson G, Nielsen J, Thorlacius H, Toth E. Capsule retention related to small bowel capsule endoscopy: a large European single-center 10-year clinical experience. United European Gastroenterol J. 2017 Aug;5(5):677-686. doi: 10.1177/2050640616675219. Epub 2016 Oct 16. PMID 28815031
- [Background] Thorndal C, Selnes O, Lei II, Koulaouzidis A. A systematic review of capsule aspiration in capsule endoscopy. Ann Transl Med. 2024 Feb 1;12(1):12. doi: 10.21037/atm-23-763. Epub 2023 Aug 28. PMID 38304904
- [Background] Mehta CR, Pocock SJ. Adaptive increase in sample size when interim results are promising: a practical guide with examples. Stat Med. 2011 Dec 10;30(28):3267-84. doi: 10.1002/sim.4102. Epub 2010 Nov 30. PMID 22105690